CLINICAL TRIAL: NCT03607799
Title: A Culturally-tailored Personalized Nutrition Intervention in South Asian Women at Risk of Gestational Diabetes Mellitus
Brief Title: A Culturally-tailored Personalized Nutrition Intervention in South Asian Women at Risk of Gestational Diabetes
Acronym: DESI-GDM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other); Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4886
Record Dates: First submitted 2018-07-12; First posted 2018-07-31 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Diabetes, Gestational
Keywords: South Asian; diet
MeSH Terms: conditions — Diabetes, Gestational | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: Human
Who Masked: Outcomes Assessor
Masking Description: Those assessing the primary and secondary clinical outcomes are masked to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Intervention (Experimental): A personalized nutrition plan will be developed for each woman and will respect faith-based food choices and regional preferences. The plan will be delivered by a culturally congruent health coach, and consider baseline dietary intake, energy balance for recommended gestational weight gain, personal values and preferences, through setting 2-4 "SMART" goals. Participants assigned to the intervention group will receive text messages. Participants assigned to the intervention group will be given a Fitbit to track their steps and will receive simple text messages weekly, aimed at increasing walking. They will be given PDF resources that provide advice on healthy eating, physical activity, and other lifestyle factors during pregnancy plus additional materials adapted specifically for the South Asian community.
  Interventions: Behavioral: Dietary Intervention
- Control (Active Comparator): Participants in the control group will receive simple text messages weekly, aimed at increasing walking. They will be given PDF resources that provide advice on healthy eating, physical activity, and other lifestyle factors during pregnancy plus additional materials adapted specifically for the South Asian community.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Dietary Intervention — Individualized diet advice will be developed for each participant by a dietitian familiar with South Asian foods.
  Arms: Dietary Intervention
Behavioral: Control — Control group participants will be provided with PDFs, website links to encourage healthy eating, physical activity, and other lifestyle factors during pregnancy. They will also receive weekly text messages aimed at increasing walking.
  Arms: Control

SUMMARY:
This trial will assess the impact of a culturally tailored, personalized nutrition intervention on glycemic response to an oral glucose load (as measured by the area-under-the curve glucose) in high-risk pregnancies of South Asian women. The intervention targets two at-risk individuals: mother and infant, "breaking the cycle" of maternal gestational dysglycemia, excess infant adiposity and insulin resistance, and CVD in both mother and baby. The findings of this study will be important in guiding future evidence-based recommendations and public health policies to manage gestational glycemia in pregnant women at risk of GDM.

DETAILED DESCRIPTION:
The DESI-GDM study is a randomized study to assess the impact of a culturally tailored, personalized nutrition intervention on glycemic response to an oral glucose load in high-risk pregnancies of South Asian women. Eligible South Asian pregnant women will be randomized to intervention or control.

South Asians (SA), people whose ancestors are from India, Pakistan, Bangladesh, or Sri Lanka, are the largest non-white ethnic group in Canada, and are at high risk of type 2 diabetes mellitus (T2DM) and early cardiovascular disease (CVD). SA women have at least double the risk of gestational diabetes (GDM) of white European women, and risk factors for future T2DM in the offspring including higher birthweight, more adipose tissue, and reduced insulin sensitivity, are more common in SA infants of mothers with GDM than infants born to mothers without GDM.

Building on our findings from the South Asian prospective birth cohort (START), which identified diet as a key modifiable risk factor for GDM, we have developed a dietary intervention. The women we spoke with expressed a desire to learn more about healthy eating to prevent diabetes during pregnancy and were keen to use mobile health technology.

The objectives of this trial among pregnant women of South Asian descent are to:

1. Evaluate the effectiveness of a culturally-tailored personalized nutrition intervention delivered by a trained health coach to improve blood sugar levels in South Asian women to a greater extant than usual dietary advice.
2. Evaluate the effectiveness of a culturally-tailored personalized nutrition intervention delivered by a trained health coach to pregnant South Asian women in the reduction of the incidence of gestational diabetes mellitus to a greater extent than usual dietary advice.

The findings of this study will be important in guiding future evidence-based recommendations and public health policies to manage gestational glycemia in pregnant women at risk of GDM.

ELIGIBILITY:
Inclusion Criteria:

* pregnant
* South Asian ancestry
* gestational week 12-18
* singleton pregnancy
* at least 2 of the following:

  1. age > 29
  2. low diet quality (assessed with a short diet questionnaire)
  3. family history of type 2 diabetes in first-degree relative
  4. gestational diabetes during a previous pregnancy
  5. pre-pregnancy body-mass-index ≥23.17

Exclusion Criteria:

* type 1 or type 2 diabetes
* high blood pressure (>140 mm Hg systolic or >90 mm Hg diastolic)
* poor understanding of English
* unwillingness to modify diet
* at high risk of adverse pregnancy outcomes other than gestational diabetes (e.g. twins or higher-order multiples, use of fertility treatment(s), pre-existing hypertension, history of placenta previa or pre-term birth)
* enrollment in another study
* does not have a smartphone
* not willing to walk
* excessive nausea and/or vomiting

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Glucose area-under-the-curve (glucose AUC) | 3 months
  A measure of glycemic response, glucose AUC is a continuous measure of the response to a 75-g oral glucose tolerance test, and is calculated by the trapezoidal method using the fasting, 1-h, and 2-h glucose.

SECONDARY OUTCOMES:
Gestational diabetes mellitus | 3 months
  Gestational diabetes mellitus is classified using the cut-offs derived in a large cohort of South Asian women from the "Born in Bradford": fasting glucose level >= 5.2 mmol/L, or 2-hour post-load level >=7.2 mmol/L.

OTHER OUTCOMES:
Maternal blood pressure | 3 months
  We measure maternal blood pressure at baseline and the OGTT visit.
Maternal pregnancy complications | 3 months
  Pregnancy complications will be noted at coaching contacts.

CONTACTS AND LOCATIONS:
Overall Officials: Russell J de Souza, ScD, Principal Investigator — McMaster University
Locations (1):
- Farah Khan, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Request for data will be assessed on a case by case basis.

REFERENCES:
- [Background] HAPO Study Cooperative Research Group; Metzger BE, Lowe LP, Dyer AR, Trimble ER, Chaovarindr U, Coustan DR, Hadden DR, McCance DR, Hod M, McIntyre HD, Oats JJ, Persson B, Rogers MS, Sacks DA. Hyperglycemia and adverse pregnancy outcomes. N Engl J Med. 2008 May 8;358(19):1991-2002. doi: 10.1056/NEJMoa0707943. PMID 18463375
- [Background] Lee AJ, Hiscock RJ, Wein P, Walker SP, Permezel M. Gestational diabetes mellitus: clinical predictors and long-term risk of developing type 2 diabetes: a retrospective cohort study using survival analysis. Diabetes Care. 2007 Apr;30(4):878-83. doi: 10.2337/dc06-1816. PMID 17392549
- [Background] Bellamy L, Casas JP, Hingorani AD, Williams D. Type 2 diabetes mellitus after gestational diabetes: a systematic review and meta-analysis. Lancet. 2009 May 23;373(9677):1773-9. doi: 10.1016/S0140-6736(09)60731-5. PMID 19465232
- [Background] Gunderson EP, Chiang V, Pletcher MJ, Jacobs DR, Quesenberry CP, Sidney S, Lewis CE. History of gestational diabetes mellitus and future risk of atherosclerosis in mid-life: the Coronary Artery Risk Development in Young Adults study. J Am Heart Assoc. 2014 Mar 12;3(2):e000490. doi: 10.1161/JAHA.113.000490. PMID 24622610
- [Background] Kim SY, Sharma AJ, Callaghan WM. Gestational diabetes and childhood obesity: what is the link? Curr Opin Obstet Gynecol. 2012 Dec;24(6):376-81. doi: 10.1097/GCO.0b013e328359f0f4. PMID 23000698
- [Background] Feig DS, Zinman B, Wang X, Hux JE. Risk of development of diabetes mellitus after diagnosis of gestational diabetes. CMAJ. 2008 Jul 29;179(3):229-34. doi: 10.1503/cmaj.080012. PMID 18663202
- [Background] Kim C, Newton KM, Knopp RH. Gestational diabetes and the incidence of type 2 diabetes: a systematic review. Diabetes Care. 2002 Oct;25(10):1862-8. doi: 10.2337/diacare.25.10.1862. PMID 12351492
- [Background] Clausen TD, Mathiesen ER, Hansen T, Pedersen O, Jensen DM, Lauenborg J, Damm P. High prevalence of type 2 diabetes and pre-diabetes in adult offspring of women with gestational diabetes mellitus or type 1 diabetes: the role of intrauterine hyperglycemia. Diabetes Care. 2008 Feb;31(2):340-6. doi: 10.2337/dc07-1596. Epub 2007 Nov 13. PMID 18000174
- [Background] Aceti A, Santhakumaran S, Logan KM, Philipps LH, Prior E, Gale C, Hyde MJ, Modi N. The diabetic pregnancy and offspring blood pressure in childhood: a systematic review and meta-analysis. Diabetologia. 2012 Nov;55(11):3114-27. doi: 10.1007/s00125-012-2689-8. Epub 2012 Sep 5. PMID 22948491
- [Background] Rana A, de Souza RJ, Kandasamy S, Lear SA, Anand SS. Cardiovascular risk among South Asians living in Canada: a systematic review and meta-analysis. CMAJ Open. 2014 Jul 22;2(3):E183-91. doi: 10.9778/cmajo.20130064. eCollection 2014 Jul. PMID 25295238
- [Background] Anand SS, Gupta M, Teo KK, Schulze KM, Desai D, Abdalla N, Zulyniak M, de Souza R, Wahi G, Shaikh M, Beyene J, de Villa E, Morrison K, McDonald SD, Gerstein H; South Asian Birth Cohort (START) - Canada Investigators. Causes and consequences of gestational diabetes in South Asians living in Canada: results from a prospective cohort study. CMAJ Open. 2017 Aug 9;5(3):E604-E611. doi: 10.9778/cmajo.20170027. PMID 28800568
- [Background] Donazar-Ezcurra M, Lopez-Del Burgo C, Bes-Rastrollo M. Primary prevention of gestational diabetes mellitus through nutritional factors: a systematic review. BMC Pregnancy Childbirth. 2017 Jan 13;17(1):30. doi: 10.1186/s12884-016-1205-4. PMID 28086820
- [Background] Tieu J, Shepherd E, Middleton P, Crowther CA. Dietary advice interventions in pregnancy for preventing gestational diabetes mellitus. Cochrane Database Syst Rev. 2017 Jan 3;1(1):CD006674. doi: 10.1002/14651858.CD006674.pub3. PMID 28046205
- [Background] Farrar D, Fairley L, Santorelli G, Tuffnell D, Sheldon TA, Wright J, van Overveld L, Lawlor DA. Association between hyperglycaemia and adverse perinatal outcomes in south Asian and white British women: analysis of data from the Born in Bradford cohort. Lancet Diabetes Endocrinol. 2015 Oct;3(10):795-804. doi: 10.1016/S2213-8587(15)00255-7. Epub 2015 Sep 6. PMID 26355010
- [Background] Mukerji G, Chiu M, Shah BR. Gestational diabetes mellitus and pregnancy outcomes among Chinese and South Asian women in Canada. J Matern Fetal Neonatal Med. 2013 Feb;26(3):279-84. doi: 10.3109/14767058.2012.735996. Epub 2012 Oct 29. PMID 23039093
- [Background] Anand SS, Vasudevan A, Gupta M, Morrison K, Kurpad A, Teo KK, Srinivasan K; START Cohort Study Investigators. Rationale and design of South Asian Birth Cohort (START): a Canada-India collaborative study. BMC Public Health. 2013 Jan 28;13:79. doi: 10.1186/1471-2458-13-79. PMID 23356884
- [Background] Lesser IA, Gasevic D, Lear SA. The association between acculturation and dietary patterns of South Asian immigrants. PLoS One. 2014 Feb 18;9(2):e88495. doi: 10.1371/journal.pone.0088495. eCollection 2014. PMID 24558396
- [Background] Simmons D, Williams R. Dietary practices among Europeans and different South Asian groups in Coventry. Br J Nutr. 1997 Jul;78(1):5-14. doi: 10.1079/bjn19970114. PMID 9292755
- [Background] Streuling I, Beyerlein A, von Kries R. Can gestational weight gain be modified by increasing physical activity and diet counseling? A meta-analysis of interventional trials. Am J Clin Nutr. 2010 Oct;92(4):678-87. doi: 10.3945/ajcn.2010.29363. Epub 2010 Jul 28. PMID 20668049
- [Background] Hui A, Back L, Ludwig S, Gardiner P, Sevenhuysen G, Dean H, Sellers E, McGavock J, Morris M, Bruce S, Murray R, Shen GX. Lifestyle intervention on diet and exercise reduced excessive gestational weight gain in pregnant women under a randomised controlled trial. BJOG. 2012 Jan;119(1):70-7. doi: 10.1111/j.1471-0528.2011.03184.x. Epub 2011 Oct 21. PMID 22017967
- [Background] Walsh JM, McGowan CA, Mahony R, Foley ME, McAuliffe FM. Low glycaemic index diet in pregnancy to prevent macrosomia (ROLO study): randomised control trial. BMJ. 2012 Aug 30;345:e5605. doi: 10.1136/bmj.e5605. PMID 22936795
- [Background] Tanentsapf I, Heitmann BL, Adegboye AR. Systematic review of clinical trials on dietary interventions to prevent excessive weight gain during pregnancy among normal weight, overweight and obese women. BMC Pregnancy Childbirth. 2011 Oct 26;11:81. doi: 10.1186/1471-2393-11-81. PMID 22029725
- [Background] Streuling I, Beyerlein A, Rosenfeld E, Hofmann H, Schulz T, von Kries R. Physical activity and gestational weight gain: a meta-analysis of intervention trials. BJOG. 2011 Feb;118(3):278-84. doi: 10.1111/j.1471-0528.2010.02801.x. Epub 2010 Dec 7. PMID 21134106
- [Background] Ronnberg AK, Nilsson K. Interventions during pregnancy to reduce excessive gestational weight gain: a systematic review assessing current clinical evidence using the Grading of Recommendations, Assessment, Development and Evaluation (GRADE) system. BJOG. 2010 Oct;117(11):1327-34. doi: 10.1111/j.1471-0528.2010.02619.x. PMID 20840691
- [Background] Ha V, Bonner AJ, Jadoo JK, Beyene J, Anand SS, de Souza RJ. The effects of various diets on glycemic outcomes during pregnancy: A systematic review and network meta-analysis. PLoS One. 2017 Aug 3;12(8):e0182095. doi: 10.1371/journal.pone.0182095. eCollection 2017. PMID 28771519
- [Background] Thangaratinam S, Rogozinska E, Jolly K, Glinkowski S, Roseboom T, Tomlinson JW, Kunz R, Mol BW, Coomarasamy A, Khan KS. Effects of interventions in pregnancy on maternal weight and obstetric outcomes: meta-analysis of randomised evidence. BMJ. 2012 May 16;344:e2088. doi: 10.1136/bmj.e2088. PMID 22596383
- [Background] Sahariah SA, Potdar RD, Gandhi M, Kehoe SH, Brown N, Sane H, Coakley PJ, Marley-Zagar E, Chopra H, Shivshankaran D, Cox VA, Jackson AA, Margetts BM, Fall CH. A Daily Snack Containing Leafy Green Vegetables, Fruit, and Milk before and during Pregnancy Prevents Gestational Diabetes in a Randomized, Controlled Trial in Mumbai, India. J Nutr. 2016 Jul;146(7):1453S-60S. doi: 10.3945/jn.115.223461. Epub 2016 Jun 8. PMID 27281802
- [Background] Edvardsson K, Ivarsson A, Eurenius E, Garvare R, Nystrom ME, Small R, Mogren I. Giving offspring a healthy start: parents' experiences of health promotion and lifestyle change during pregnancy and early parenthood. BMC Public Health. 2011 Dec 15;11:936. doi: 10.1186/1471-2458-11-936. PMID 22171644
- [Background] Devine CM, Bove CF, Olson CM. Continuity and change in women's weight orientations and lifestyle practices through pregnancy and the postpartum period: the influence of life course trajectories and transitional events. Soc Sci Med. 2000 Feb;50(4):567-82. doi: 10.1016/s0277-9536(99)00314-7. PMID 10641808
- [Background] Greenhalgh T, Clinch M, Afsar N, Choudhury Y, Sudra R, Campbell-Richards D, Claydon A, Hitman GA, Hanson P, Finer S. Socio-cultural influences on the behaviour of South Asian women with diabetes in pregnancy: qualitative study using a multi-level theoretical approach. BMC Med. 2015 May 21;13:120. doi: 10.1186/s12916-015-0360-1. PMID 25998551
- [Background] Subar AF, Kirkpatrick SI, Mittl B, Zimmerman TP, Thompson FE, Bingley C, Willis G, Islam NG, Baranowski T, McNutt S, Potischman N. The Automated Self-Administered 24-hour dietary recall (ASA24): a resource for researchers, clinicians, and educators from the National Cancer Institute. J Acad Nutr Diet. 2012 Aug;112(8):1134-7. doi: 10.1016/j.jand.2012.04.016. Epub 2012 Jun 15. No abstract available. PMID 22704899
- [Background] Khan SA, Jackson RT, Momen B. The Relationship between Diet Quality and Acculturation of Immigrated South Asian American Adults and Their Association with Metabolic Syndrome. PLoS One. 2016 Jun 14;11(6):e0156851. doi: 10.1371/journal.pone.0156851. eCollection 2016. PMID 27299862
- [Background] Anand SS, Samaan Z, Middleton C, Irvine J, Desai D, Schulze KM, Sothiratnam S, Hussain F, Shah BR, Pare G, Beyene J, Lear SA; South Asian Heart Risk Assessment Investigators. A Digital Health Intervention to Lower Cardiovascular Risk: A Randomized Clinical Trial. JAMA Cardiol. 2016 Aug 1;1(5):601-6. doi: 10.1001/jamacardio.2016.1035. PMID 27438754
- [Background] Samaan Z, Schulze KM, Middleton C, Irvine J, Joseph P, Mente A, Shah BR, Pare G, Desai D, Anand SS; SAHARA Investigators. South Asian Heart Risk Assessment (SAHARA): Randomized Controlled Trial Design and Pilot Study. JMIR Res Protoc. 2013 Aug 20;2(2):e33. doi: 10.2196/resprot.2621. PMID 23965279
- [Background] Anand SS, Gupta MK, Schulze KM, Desai D, Abdalla N, Wahi G, Wade C, Scheufler P, McDonald SD, Morrison KM, Vasudevan A, Dwarakanath P, Srinivasan K, Kurpad A, Gerstein HC, Teo KK. What accounts for ethnic differences in newborn skinfold thickness comparing South Asians and White Caucasians? Findings from the START and FAMILY Birth Cohorts. Int J Obes (Lond). 2016 Feb;40(2):239-44. doi: 10.1038/ijo.2015.171. Epub 2015 Aug 28. PMID 26315840
- [Background] Chow CK, Redfern J, Hillis GS, Thakkar J, Santo K, Hackett ML, Jan S, Graves N, de Keizer L, Barry T, Bompoint S, Stepien S, Whittaker R, Rodgers A, Thiagalingam A. Effect of Lifestyle-Focused Text Messaging on Risk Factor Modification in Patients With Coronary Heart Disease: A Randomized Clinical Trial. JAMA. 2015 Sep 22-29;314(12):1255-63. doi: 10.1001/jama.2015.10945. PMID 26393848
- [Background] Pludwinski S, Ahmad F, Wayne N, Ritvo P. Participant experiences in a smartphone-based health coaching intervention for type 2 diabetes: A qualitative inquiry. J Telemed Telecare. 2016 Apr;22(3):172-8. doi: 10.1177/1357633X15595178. Epub 2015 Jul 21. PMID 26199275
- [Background] Canadian Diabetes Association Clinical Practice Guidelines Expert Committee; Cheng AY. Canadian Diabetes Association 2013 clinical practice guidelines for the prevention and management of diabetes in Canada. Introduction. Can J Diabetes. 2013 Apr;37 Suppl 1:S1-3. doi: 10.1016/j.jcjd.2013.01.009. Epub 2013 Mar 26. No abstract available. PMID 24070926
- [Background] Mohan V, Mahalakshmi MM, Bhavadharini B, Maheswari K, Kalaiyarasi G, Anjana RM, Uma R, Usha S, Deepa M, Unnikrishnan R, Pastakia SD, Malanda B, Belton A, Kayal A. Comparison of screening for gestational diabetes mellitus by oral glucose tolerance tests done in the non-fasting (random) and fasting states. Acta Diabetol. 2014 Dec;51(6):1007-13. doi: 10.1007/s00592-014-0660-5. Epub 2014 Oct 15. PMID 25315629
- [Background] Sen B, Bose K, Shaikh S, Mahalanabis D. Prediction equations for body-fat percentage in Indian infants and young children using skinfold thickness and mid-arm circumference. J Health Popul Nutr. 2010 Jun;28(3):221-9. doi: 10.3329/jhpn.v28i3.5548. PMID 20635632
- [Background] Luoto R, Kinnunen TI, Aittasalo M, Kolu P, Raitanen J, Ojala K, Mansikkamaki K, Lamberg S, Vasankari T, Komulainen T, Tulokas S. Primary prevention of gestational diabetes mellitus and large-for-gestational-age newborns by lifestyle counseling: a cluster-randomized controlled trial. PLoS Med. 2011 May;8(5):e1001036. doi: 10.1371/journal.pmed.1001036. Epub 2011 May 17. PMID 21610860
- [Background] Poston L, Bell R, Croker H, Flynn AC, Godfrey KM, Goff L, Hayes L, Khazaezadeh N, Nelson SM, Oteng-Ntim E, Pasupathy D, Patel N, Robson SC, Sandall J, Sanders TA, Sattar N, Seed PT, Wardle J, Whitworth MK, Briley AL; UPBEAT Trial Consortium. Effect of a behavioural intervention in obese pregnant women (the UPBEAT study): a multicentre, randomised controlled trial. Lancet Diabetes Endocrinol. 2015 Oct;3(10):767-77. doi: 10.1016/S2213-8587(15)00227-2. Epub 2015 Jul 9. PMID 26165396
- [Background] Quinlivan JA, Lam LT, Fisher J. A randomised trial of a four-step multidisciplinary approach to the antenatal care of obese pregnant women. Aust N Z J Obstet Gynaecol. 2011 Apr;51(2):141-6. doi: 10.1111/j.1479-828X.2010.01268.x. Epub 2011 Jan 31. PMID 21466516
- [Background] Koivusalo SB, Rono K, Klemetti MM, Roine RP, Lindstrom J, Erkkola M, Kaaja RJ, Poyhonen-Alho M, Tiitinen A, Huvinen E, Andersson S, Laivuori H, Valkama A, Meinila J, Kautiainen H, Eriksson JG, Stach-Lempinen B. Gestational Diabetes Mellitus Can Be Prevented by Lifestyle Intervention: The Finnish Gestational Diabetes Prevention Study (RADIEL): A Randomized Controlled Trial. Diabetes Care. 2016 Jan;39(1):24-30. doi: 10.2337/dc15-0511. Epub 2015 Jul 29. PMID 26223239
- [Background] Simmons D, Jelsma JG, Galjaard S, Devlieger R, van Assche A, Jans G, Corcoy R, Adelantado JM, Dunne F, Desoye G, Harreiter J, Kautzky-Willer A, Damm P, Mathiesen ER, Jensen DM, Andersen LL, Lapolla A, Dalfra M, Bertolotto A, Wender-Ozegowska E, Zawiejska A, Hill D, Rebollo P, Snoek FJ, van Poppel MN. Results From a European Multicenter Randomized Trial of Physical Activity and/or Healthy Eating to Reduce the Risk of Gestational Diabetes Mellitus: The DALI Lifestyle Pilot. Diabetes Care. 2015 Sep;38(9):1650-6. doi: 10.2337/dc15-0360. Epub 2015 Jun 25. PMID 26112044
- [Background] The Social Planning Council of Peel. An exploratory study of diabetes among South Asians in Peel. Peel, ON, 2015.
- [Background] Morency J-D, Malenfant EC, MacIssac S. Immigration and Diversity: Population Projections for Canada and its Regions, 2011 to 2036. Ottawa, ON: Statistics Canada;2017.
- [Background] Allison DB, Paultre F, Maggio C, Mezzitis N, Pi-Sunyer FX. The use of areas under curves in diabetes research. Diabetes Care. 1995 Feb;18(2):245-50. doi: 10.2337/diacare.18.2.245. PMID 7729306
- [Background] Sakaguchi K, Takeda K, Maeda M, Ogawa W, Sato T, Okada S, Ohnishi Y, Nakajima H, Kashiwagi A. Glucose area under the curve during oral glucose tolerance test as an index of glucose intolerance. Diabetol Int. 2015 May 14;7(1):53-58. doi: 10.1007/s13340-015-0212-4. eCollection 2016 Mar. PMID 30603243
- [Background] Canadian Diabetes Association Clinical Practice Guidelines Expert Committee; Thompson D, Berger H, Feig D, Gagnon R, Kader T, Keely E, Kozak S, Ryan E, Sermer M, Vinokuroff C. Diabetes and pregnancy. Can J Diabetes. 2013 Apr;37 Suppl 1:S168-83. doi: 10.1016/j.jcjd.2013.01.044. Epub 2013 Mar 26. No abstract available. PMID 24070943
- [Background] Feig DS, Berger H, Donovan L, Godbout A, Kader T, Keely E, Sanghera R. Erratum to "Diabetes and Pregnancy": Canadian Journal of Diabetes 2018;42(S1):S255-S282. Can J Diabetes. 2018 Jun;42(3):337. doi: 10.1016/j.jcjd.2018.04.006. No abstract available. PMID 29857812
- [Background] Duran A, Saenz S, Torrejon MJ, Bordiu E, Del Valle L, Galindo M, Perez N, Herraiz MA, Izquierdo N, Rubio MA, Runkle I, Perez-Ferre N, Cusihuallpa I, Jimenez S, Garcia de la Torre N, Fernandez MD, Montanez C, Familiar C, Calle-Pascual AL. Introduction of IADPSG criteria for the screening and diagnosis of gestational diabetes mellitus results in improved pregnancy outcomes at a lower cost in a large cohort of pregnant women: the St. Carlos Gestational Diabetes Study. Diabetes Care. 2014 Sep;37(9):2442-50. doi: 10.2337/dc14-0179. Epub 2014 Jun 19. PMID 24947793
- [Background] Lapolla A, Dalfra MG, Ragazzi E, De Cata AP, Fedele D. New International Association of the Diabetes and Pregnancy Study Groups (IADPSG) recommendations for diagnosing gestational diabetes compared with former criteria: a retrospective study on pregnancy outcome. Diabet Med. 2011 Sep;28(9):1074-7. doi: 10.1111/j.1464-5491.2011.03351.x. PMID 21658125
- [Background] Mission JF, Ohno MS, Cheng YW, Caughey AB. Gestational diabetes screening with the new IADPSG guidelines: a cost-effectiveness analysis. Am J Obstet Gynecol. 2012 Oct;207(4):326.e1-9. doi: 10.1016/j.ajog.2012.06.048. Epub 2012 Jun 29. PMID 22840972
- [Background] Archambault C, Arel R, Filion KB. Gestational diabetes and risk of cardiovascular disease: a scoping review. Open Med. 2014 Jan 7;8(1):e1-9. eCollection 2014. PMID 25009679
- [Derived] Stennett RN, Adamo KB, Anand SS, Bajaj HS, Bangdiwala SI, Desai D, Gerstein HC, Kandasamy S, Khan F, Lear SA, McDonald SD, Pocsai T, Ritvo P, Rogge A, Schulze KM, Sherifali D, Stearns JC, Wahi G, Williams NC, Zulyniak MA, de Souza RJ. A culturally tailored personaliseD nutrition intErvention in South ASIan women at risk of Gestational Diabetes Mellitus (DESI-GDM): a randomised controlled trial protocol. BMJ Open. 2023 May 2;13(5):e072353. doi: 10.1136/bmjopen-2023-072353. PMID 37130668

DOCUMENTS (2):
  • Study Protocol (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/99/NCT03607799/Prot_000.pdf
  • Informed Consent Form (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/99/NCT03607799/ICF_001.pdf